CLINICAL TRIAL: NCT03867968
Title: Brain Injury Support and Strategies for Families Impacted by Childhood TBI
Brief Title: Traumatic Brain Injury Positive Strategies
Acronym: TIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R44HD059255 (NIH); 5R44HD059255-04 (NIH)
Record Dates: First submitted 2019-01-17; First posted 2019-03-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIPS Intervention (Experimental): The Traumatic Brain Injury Positive Strategies (TIPS) program, is a comprehensive educational and training resource to help families. The web-based product will include: (a) the Training Center, which will provide training in a range of evidence-based strategies within a problem-solving framework; and (b) the TBI Resource Center, an extensive library of educational materials, information, and resources about childhood TBI.
  Interventions: Behavioral: TIPS Intervention
- Control (Active Comparator): An existing website related to traumatic brain injury.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: TIPS Intervention — Web-based training for family member.
  Arms: TIPS Intervention
Behavioral: Control — Traumatic Brain Injury website for family members.
  Arms: Control

SUMMARY:
This study evaluates the effectiveness of The Traumatic Brain Injury Positive Strategies (TIPS) program, a comprehensive educational and training resource to help families improve their knowledge and skills in supporting a child with TBI experiencing cognitive, behavioral, and social challenges. The application provides training in evidence-based support strategies with the goal of improving outcomes for children with TBI and their families. Half the participants will receive access to the TIPS program, while the other half will receive access to a different TBI related website.

DETAILED DESCRIPTION:
Due to the chronic nature of cognitive and behavioral problems related to TBI, parents and other family caregivers need information, resources, and training in evidence-based strategies to manage the varied and changing concerns following their child's injury. Recent research provides evidence that theory-driven, self-directed online parent training is effective in improving both child and parent outcomes.

The objective of this project is to produce the Traumatic Brain Injury Positive Strategies (TIPS) program, a comprehensive educational and training resource to help families improve their knowledge and skills to address cognitive, behavioral, and social challenges following pediatric TBI. The TIPS program will be grounded in the theory of planned behavior, which postulates that training in problem-solving leads to improved skills and increases in perceived behavioral control that mediate direct changes in parenting behaviors and indirect changes in child outcomes. The web-based product will include: (a) the Training Center, which will provide training in a range of evidence-based strategies within a problem-solving framework; and (b) the TBI Resource Center, an extensive library of educational materials, information, and resources about childhood TBI.

Approximately 216 family members will participate in the evaluation phase of this study. Participants will be randomly assigned to one of two conditions: (a) treatment (TIPS program ) or (b) control (brain injury website).

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years old or older
* Have a child age 3-18 that was hospitalized overnight with a traumatic brain injury (TBI).
* Involved in the care and support of the child with the TBI.
* Live in the same household as child with a TBI.
* The child with the TBI is able to follow simple instructions such as "please eat your toast."

Exclusion Criteria:

* Does not speak and read English.
* Does not have high speed Internet access.
* Not US resident

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
TIPS Change in Knowledge Survey | Baseline , at intervention completion an average of 4 weeks, and for a 3 month follow up after completed intervention.
  Survey to assess change in knowledge of research-based cognitive, behavioral, and social support strategies and self-efficacy about using those strategies in home and community settings.
PedsQL Family Impact | Baseline and for a 3 month follow up after completed intervention.
  Administered to measure change in impact of pediatric acute and chronic health conditions on parents and the family.
Caregiver Self-Efficacy Scale | Baseline, at intervention completion an average of 4 weeks, and for a 3 month follow up after completed intervention.
  25-question self-report measure, administered to measure the change in how comfortable caregivers feel about selected aspects of their parenting skills such as managing their child's behavior, being an advocate for their child, and dealing with school-related issues.

SECONDARY OUTCOMES:
The Pediatric Quality of Life Inventory (PedsQL) | Baseline
  23 items measuring physical, emotional, social, and school function. Caregiver report forms have been developed for children 2-18 years. The PedsQL has been used in pediatric TBI as a quality of life outcome.
PedsQL Cognitive Function | Baseline
  Measures cognitive functioning in patients with acute and chronic health conditions as well as healthy school and community populations.
Health Behavior Inventory (HBI) | Baseline, at intervention completion an average of 4 weeks, and for a 3 month follow up after completed intervention.
  20 items measuring the change in frequency of common brain injury symptoms (somatic, cognitive, and emotional). It will also be used to examine the effectiveness of the interventions in promoting symptom reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Glang, PhD, Principal Investigator — University of Oregon
Locations (1):
- Center on Brain Injury Research and Training / University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karns CM, Wade SL, Slocumb J, Keating T, Gau JM, Slomine BS, Suskauer SJ, Glang A. Traumatic Brain Injury Positive Strategies for Families: A Pilot Randomized Controlled Trial of an Online Parent-Training Program. Arch Phys Med Rehabil. 2023 Jul;104(7):1026-1034. doi: 10.1016/j.apmr.2023.03.013. Epub 2023 May 2. PMID 37142177